CLINICAL TRIAL: NCT05127239
Title: Constructing a Care Model Combing Smartphone Application to Improve Obstructive Apnea in Obesity Adults: a Longitudinal Study
Brief Title: The Effectiveness of Smartphone Application on the Serevity of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hsu Hsiu-Chin, Associate professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 201802318B0A3
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; home portable sleep monitor; smartphone application; lifestyle modification intervention
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistant who assisted in the production of serial numbers was not involved in recruitment, intervention, or data collection. In addition, the researcher who performed the data analysis did not participate in recruitment, intervention or data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- smartphone application with education (Experimental): participants were provides 3 times lifestyle modification education and using smartphone app program
  Interventions: Behavioral: Smartphone Application with lifestyle modification Intervention
- smartphone application (Experimental): participants were only provided smartphone app program
  Interventions: Behavioral: Smartphone Application with lifestyle modification Intervention
- waiting list (No Intervention): No intervention was provided, but researchers explained the results of OSA screening for participants after every examination

INTERVENTIONS:
Behavioral: Smartphone Application with lifestyle modification Intervention — The study will introduce a health-promoting lifestyle through the combination of a smartphone app (MyFitnessPal) for the experimental group, emphasizing the use of behavior change techniques to reduce weight, thereby improving the obstructive sleep apnea with overweight and obese employees in the workplace. The self-monitoring, instant feedback, and social support, as well as individualized tailor-made functions are used in intervention programs. The intervention process adopts a healthy weight reduction plan, focusing on a balanced diet, moderately reducing the calories of the food, and combining weight loss methods such as increasing exercise as the main axis, emphasizing the concept of self-monitoring of weight, calorie intake, and exercise .
  Arms: smartphone application; smartphone application with education

SUMMARY:
A two-year study design is formulated. The overall aim of this study is to examine the effectiveness of the care model combing smartphone application on improve obstructive apnea in obesity adults.

DETAILED DESCRIPTION:
This study was the second year.The purpose of this study is to evaluate the effectiveness of the lifestyle modification intervention for overweight employees with obstructive sleep apnea. A randomized control trial with single blind will be used. Stratified with proportional randomized sampling will be employed and 160 suitable participants will be recruited from 4 electronics industries in northern of Taiwan. The subjects will be randomly divided into three groups. The total duration of intervention program is 6 months. Only the intervention group received the Combining Smartphone Application with lifestyle modification Intervention. The home portable sleep monitor will be used to collect the change of AHI at baseline, 3, and 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria: a) >21 years old; b) )BMI greater than24 kg/m2; (c) the absence of any mental disorder, alcohol and drug addiction, and serious disease, such as cancer or cardiorespiratory failure; and d) Screening for OSA , AHI>5 and voluntary participation.

-

Exclusion Criteria:

* a) diagnosis of OSA and currently under treatment and；b) diagnosis of severe depression (c) have cardiopulmonary diseases and are not suitable for activities; and d) plan to become pregnant during or within 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | one night
  using the Portable sleep monitor to examine the change of Apnea-Hypopnea Index

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chin Hsu, e-mail, Principal Investigator — Department of Graduate Institute of Health Care, Chang Gung University of Science and Technology
Locations (1):
- Phison Electronics Corp, Miaoli, Taiwan